CLINICAL TRIAL: NCT06556121
Title: The Addition of a Saddle Block With Intrathecal Morphine for Analgesia in Transgender Patients Undergoing Penile Inversion Vaginoplasty: A Randomized Double-blind Placebo-controlled Trial
Brief Title: Saddle Block With IT Morphine for Penile Inversion Vaginoplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-0061-B
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Pain, Postoperative
Keywords: Saddle block; transition; pudendal nerve block; gender confirmation surgery; penile inversion Vaginoplasty
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized, parallel-group, double-blind
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patient, anesthesiologist in the operating room
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saddle block with intrathecal morphine Group (Experimental): Patients will receive a multimodal analgesic regimen with acetaminophen, NSAIDs and opioids plus a surgeon-administered pudendal nerve block by anatomical landmarks with 50mL of Normal Saline, 30mL of 0.25% Bupivacaine with epinephrine 1:200.000 and 20mL Lidocaine 1%. A volume of 20 mL of this mixture is used for the pudendal nerve block, and infiltration of the surgical incision and bilateral spermatic cord block is performed with an additional 20 mL of the same mixture of local anesthetic. 30ml of the solution is used to soak the vaginal plug made of gauze that is put inside the vaginal canal by the end of the procedure.
  Patients who are randomized to the saddle block with intrathecal morphine will receive an injection of 5mg of heavy Bupivacaine 0.75% plus 100mcg of morphine injected in the intrathecal space.
  Interventions: Procedure: Saddle block; Procedure: pudendal nerve block
- Control Group (Sham Comparator): As part of the analgesic plan, all patients will receive a multimodal analgesic regimen with acetaminophen, NSAIDs and opioids plus a surgeon-administered pudendal nerve block by anatomical landmarks with 50mL of Normal Saline, 30mL of 0.25% Bupivacaine with epinephrine 1:200.000 and 20mL Lidocaine 1%. A volume of 20 mL of this mixture is used for the pudendal nerve block, and infiltration of the surgical incision and bilateral spermatic cord block is performed with an additional 20 mL of the same mixture of local anesthetic. 30ml of the solution is used to soak the vaginal plug made of gauze that is put inside the vaginal canal by the end of the procedure.
  Patients in this group will receive a non-invasive sham saddle block in addition to the care standard.
  Interventions: Procedure: pudendal nerve block

INTERVENTIONS:
Procedure: Saddle block — The injected solution will be comprised of 5mg of heavy Bupivacaine 0.75% plus 100mcg of Morphine will be injected into the intrathecal space.
  Arms: Saddle block with intrathecal morphine Group
Procedure: pudendal nerve block — As part of the analgesic plan, all patients will receive a multimodal analgesic regimen with acetaminophen, NSAIDs and opioids plus a surgeon-administered pudendal nerve block by anatomical landmarks with a mixture of Local Anesthetic as follows: 50mL of Normal Saline, 30mL of 0.25% Bupivacaine with epinephrine 1:200.000 and 20mL Lidocaine 1%. A volume of 20 mL of this mixture is used for the pudendal nerve block, and infiltration of the surgical incision and bilateral spermatic cord block is performed with an additional 20 mL of the same mixture of local anesthetic. 30ml of the solution is used to soak the vaginal plug made of gauze that is put inside the vaginal canal by the end of the procedure.

SUMMARY:
Penile Inversion Vaginoplasty (PIV) is a transition-related surgery (TRS) that is associated with severe postoperative pain. The optimal pain management strategies for this surgery remain unknown. We hypothesized that the addition of a saddle block with intrathecal morphine would yield clinically important analgesic benefits.

DETAILED DESCRIPTION:
PIV is a TRS offered for male-to-female transition associated with severe postoperative pain despite contemporary analgesic strategies, including opioid-based multimodal systemic analgesia and local anesthetic-based pudendal nerve block. Intrathecal opioids directly target the nociceptors in the spinal cord and can provide potent analgesia for abdominopelvic procedures, including PIV, but are associated with important dose-related adverse effects with rostral spread within the cerebrospinal fluid.

Motor-sparing saddle block using ultra-low dose hyperbaric spinal anesthesia has been successfully implemented as the standard of care for anesthesia in patients undergoing ambulatory perianal procedures at WCH. Saddle block produces reliable sensory anesthesia and long-lasting analgesia of the perineum ("saddle") as the hyperbaric local anesthetic preferentially blocks the small pain fibers of the sacral nerve roots with gravity when the patient is placed in the seated position. With the aim to directly target the opioid nociceptors in the sacral roots and limit rostral opioid spread (and associated opioid-related adverse effects), we recently began to offer a presurgical saddle block with a low dose of intrathecal morphine (100mcg) to patients undergoing PIV at WCH with excellent anecdotal results. Therefore, we are undertaking the present randomized placebo-controlled study to determine whether or not the addition of a saddle block with IT morphine to multimodal systemic analgesia and surgeon-administered pudendal nerve block provides superior analgesia to multimodal systemic analgesia and surgeon-administered pudendal nerve block alone.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients
* Ages 18-70 years
* Penile Inversion Vaginoplasty

Exclusion Criteria:

* Local infection
* History of use of over 30mg oxycodone or equivalent per day.
* Contraindication to a component of multi-modal analgesia
* Complications or adverse events unrelated to the local anesthetic that precludes evaluation of the primary and secondary outcome measures.
* Unable to speak or read English.
* Revision and Vulvaplasty surgeries

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male-to-female transitioning patient
Enrollment: 40 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid (analgesic) consumption | 48 hours
  Consumption intra-operatively, total in-hospital postoperative consumption measured oral morphine equivalents (MEQ)

SECONDARY OUTCOMES:
Time to first analgesic request | 24 hours
  At recovery room discharge and hospital discharge
Pain Assessment (VAS) | Up to 48 hours post-operatively
  Visual Analogue Scale(VAS) - Pain:Overall pain assessed at rest and on movement A continuous scale comprised of a 100mm (10cm) horizontal line, anchored by 2 verbal descriptions No Pain to Worst Pain
Incidence of opioid-related side effects | Up to 48 hours post-operatively
  Itching, respiratory depression, hypotension, nausea and vomiting
Presence of Block-related complications | Up to 48 hours post-operatively
  Persistent paresthesia, post dural puncture headache
Quality of Life scores | 48 hours post-operatively
  Quality of Recovery (QR15) scores at 48 hours will be the second primary outcome.
  QR15 is a measurement of quality of recovery after surgery and anesthesia that has been psychometrically tested and validated. Reporting of outcome measures on a scale of 0 to 10 (0=None of the time and 10=All of the time). There are a total of 40 items/questions.
Patient Satisfaction with Analgesic Technique and Pain management | 24 hours post-operatively
  A Patient Diary will be completed to assess overall satisfaction with analgesic technique

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD, Principal Investigator — Women's College Hospital; Laura Giron-Arango, MD, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swisher MW, Dolendo IM, Sztain JF, Alexander BS, Tsuda PS, Anger JT, Said ET. Intrathecal Morphine Injection for Postoperative Analgesia Following Gender-Affirming Pelvic Surgery: A Retrospective Case-Control Study. Cureus. 2023 Mar 27;15(3):e36748. doi: 10.7759/cureus.36748. eCollection 2023 Mar. PMID 37123779
- [Background] Yung EM, Abdallah FW, Todaro C, Spence E, Grant A, Brull R. Optimal local anesthetic regimen for saddle block in ambulatory anorectal surgery: an evidence-based systematic review. Reg Anesth Pain Med. 2020 Sep;45(9):733-739. doi: 10.1136/rapm-2020-101603. Epub 2020 Jul 22. PMID 32699103
- [Background] Hein A, Rosblad P, Gillis-Haegerstrand C, Schedvins K, Jakobsson J, Dahlgren G. Low dose intrathecal morphine effects on post-hysterectomy pain: a randomized placebo-controlled study. Acta Anaesthesiol Scand. 2012 Jan;56(1):102-9. doi: 10.1111/j.1399-6576.2011.02574.x. PMID 22150410
- [Background] DI Filippo A, Capezzuoli T, Fambrini M, Cariti G, Orlandi G, Vannucci G, Borracci T, DI Nallo L, Mazzella M, Petraglia F. Enhanced recovery after gynecological surgery: comparison between intrathecal and intravenous morphine multimodal analgesia. Minerva Obstet Gynecol. 2023 Apr;75(2):145-149. doi: 10.23736/S2724-606X.21.04961-7. Epub 2021 Dec 1. PMID 34851074
- [Background] Shim JW, Cho YJ, Moon HW, Park J, Lee HM, Kim YS, Moon YE, Hong SH, Chae MS. Analgesic efficacy of intrathecal morphine and bupivacaine during the early postoperative period in patients who underwent robotic-assisted laparoscopic prostatectomy: a prospective randomized controlled study. BMC Urol. 2021 Feb 26;21(1):30. doi: 10.1186/s12894-021-00798-4. PMID 33637066
- [Background] Chin P, Yuan N, Zaliznyak M, Stelmar J, Garcia M. Effectiveness of Pudendal Nerve Blocks on Postoperative Pain Control and Reduction in Opioid Usage after Gender-affirming Vaginoplasty. The Journal of Sexual Medicine. 2022;19(4, Supplement 1):S79. doi:10.1016/j.jsxm.2022.01.166